CLINICAL TRIAL: NCT02803658
Title: Impact of Male Smoking on the Couple's Infertility: Two-centre Case-control Study
Brief Title: Impact of Male Smoking on the Couple's Infertility
Acronym: TABAFERTIMASC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PHRCIR09-DR-DEVAUX-MME
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Infertility
Keywords: smoking
MeSH Terms: conditions — Infertility; Smoking

ARMS (2):
- infertile couples (Experimental): smoking behavior
  Interventions: Behavioral: smoking behavior; Biological: Sperm collection
- Fertile couples (Active Comparator): smoking behavior
  Interventions: Behavioral: smoking behavior

INTERVENTIONS:
Behavioral: smoking behavior
Biological: Sperm collection
  Arms: infertile couples

SUMMARY:
About 15% of couples consult for difficulties achieving pregnancy. In about two-thirds of cases, a male component is identified, but is not always sufficient to explain infertility. In the majority of cases, the cause cannot be clearly identified and multiple abnormalities may be detected in both partners.

Many factors concerning lifestyle and environment (medications, alcohol, smoking, pollution, exposure to heat, toxins, xenobiotic oestrogens, etc.) may impact on fertility. These factors may also impact on the fertility of the children conceived, which is described as an intergenerational effect (alteration of the fertility of boys exposed to smoking in utero).

Few scientific studies with a high level of proof have been published on the impact of smoking on the couple's fertility. Gonadal functioning and the quality of gametes can be altered by these environmental factors, which may trigger a process of apoptosis or alteration of the DNA of gametes (sperm DNA fragmentation). Other modifications include DNA methylation and histone acetylation, which control gene expression and are grouped under the term epigenetic modifications. More recently, oestrogens has been shown to be involved in male reproductive function by acting on spermatogenesis, spermiogenesis and epididymal maturation. Demonstration of an active aromatase (Arom) (mRNA, protein and activity) in ejaculated human spermatozoa suggests the synthesis of small quantities of oestrogens in spermatozoa. The study of transcript profiles could provide information about the quality of spermatogenesis and/or spermiogenesis and during the first steps of embryonic development. Confocal microscopy has colocalized the aromatase on the head, midpiece and tail and can be used to assess the quality of the acrosome with anti-CD-46 monoclonal antibody. Even low concentrations of xenobiotic oestrogens can exert biological effects on certain functions of murine or human spermatozoa, accelerating capacitation and the acrosome reaction. These factors are all the more effective when they act in combination, as human gametes appear to be more sensitive to their action than murine gametes All studies conducted to date have investigated the impact of toxins either on one of the partners or in the children born to the couple. No detailed and high-level scientific study has studied both partners and the quality of their embryos.

DETAILED DESCRIPTION:
The Amiens University Hospital Cytogenetic, CECOS Reproduction Biology, and the assisted reproductive technology departments in collaboration with Caen University Hospital (members of G4) want to conduct this type of routine clinical practice follow-up study in the context of an inter-regional research grant (PHRC). These 2 University Hospitals are situated in agricultural regions with potential polluting industries. The recruitment of these centres comprises younger couples presenting with infertility for which a cause cannot always be demonstrated and in which the percentage of ART by ICSI is higher than the national average (close to 75% vs 60%). This population also presents a higher cancer risk than in other regions.

This research project concerns evaluation of the impact of male smoking on the couple's fertility and will consist of a two-centre case-control study.

ELIGIBILITY:
Inclusion Criteria:

* Fertile couples = control cases (with spontaneously conceived a child with a time required to design less than 12 months) and whose wife gives birth in one of the two maternity hospitals participating in the study
* All couples candidates for AMP: reproductive age couples (Female age <35 years of age men <40 years), infertility (primary infertility, inability to conceive after 12 months of no sex protected). 1st or 2nd attempt at in vitro fertilization
* For infertile couples, couples in which we note

  1. spouses have sperm characteristics compatible with a natural pregnancy: an normospermie (> 20 million / ml) or moderate oligozoospermia (5-20 million sperm per ml) idiopathic (or exclusion criteria)
  2. where the partner does not exhibit anovulation or tubal pathology-proven utero, whose ovarian reserve is normal (FSH and estradiol rate J2 / 3 of cycle) ,.

Exclusion Criteria:

* Female age > 35 years Women> 45 years
* Co- infections of one of the two members of the couple (or 2) by HIV, HBV and / or HCV
* Severe Oligospermia humans ( <5000 000 sperm) or azzoospermie
* A normospermie or moderate oligozoospermia (5-20 million sperm per ml) nonidiopathic
* Will also be excluded couples where the partner has anovulation or uterotubal proven pathology , impaired ovarian reserve or chronic viral disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Carbon monoxide | 3 months
  in expired air using CO-tester®
Cotinine rate (micromol/L) | 3 months
  quantitative dosages of blood and / or seminal fluid or in the hair

CONTACTS AND LOCATIONS:
Overall Officials: Aviva DEVAUX, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - CHU Caen, Caen